CLINICAL TRIAL: NCT06709547
Title: Which Trauma Severity Score (ISS, NISS, RTS, or TRISS) Best Predicts Mortality in Trauma Patients? A Prospective Observational Study
Brief Title: Mortality Prediction Using Trauma Scores
Status: Recruiting | Type: Observational
Sponsor: Al-Nahrain University (Other)
Responsible Party: Principal Investigator, Abdul-Ilah R. Khamis, Principal Investigator, Al-Nahrain University
Other Study IDs: UNCOMIRB20241123
Record Dates: First submitted 2024-11-23; First posted 2024-11-29 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Trauma, Multiple
Keywords: ISS; NISS; RTS; TISS
MeSH Terms: conditions — Multiple Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of this prospective cohort study is to compare the predictive utility of the Injury Severity Score (ISS), New Injury Severity Score (NISS), Revised Trauma Score (RTS), and Trauma and Injury Severity Score (TRISS) in determining mortality outcomes among trauma patients admitted to the trauma and emergency department at Kadhimiya Educational Hospital in Baghdad.

The main questions it aims to answer are:

Which trauma scoring system provides the most accurate prediction of mortality? Are there specific trauma patient subgroups where one scoring system outperforms the others?

Participants will:

Be assessed using all four trauma scoring systems (ISS, NISS, RTS, and TRISS) upon admission to the trauma and emergency department.

Have their clinical outcomes, including mortality, length of hospital stay, ICU admission, and discharge status, monitored throughout their hospital stay to evaluate the accuracy and utility of each scoring system in predicting patient outcomes.

DETAILED DESCRIPTION:
Trauma remains a leading cause of morbidity and mortality worldwide, with millions of individuals affected annually. The severity of trauma injuries can vary widely, ranging from minor to life-threatening, and effective management often hinges on the ability to quickly assess the severity of injury and predict patient outcomes, including mortality. Accurate and timely prognostication is essential for prioritizing care, guiding treatment decisions, and allocating resources in trauma care settings. Trauma severity scoring systems have been developed to assist in these assessments, with the most commonly used being the Injury Severity Score (ISS), the New Injury Severity Score (NISS), the Revised Trauma Score (RTS), and the Trauma and Injury.

Injury Severity Score (ISS) The Injury Severity Score (ISS) was developed in the 1970s as a way to quantify the severity of trauma-related injuries based on anatomic regions of injury. The ISS assigns scores to the most severe injuries in six body regions, and the sum of the squares of the highest AIS (abbreviated Injury Score) from each of the three most severely injured regions determines the total score. ISS is widely used for risk stratification in trauma patients and has been validated as a predictor of mortality in various populations.

New Injury Severity Score (NISS) The New Injury Severity Score (NISS), introduced in the 1990s, improves upon the ISS by utilizing the three most severe injuries across any body region rather than restricting it to the highest injuries from three predefined regions. Research has shown that NISS is more predictive of mortality than ISS, particularly in patients with polytrauma or multiple severe injuries across different body regions. Despite its advantages, Revised Trauma Score (RTS) The Revised Trauma Score (RTS) is a physiological scoring system based on three clinical parameters: Glasgow Coma Scale (GCS), systolic blood pressure (SBP), and respiratory rate (RR). Unlike ISS and NISS, RTS focuses on the immediate physiological status of the patient rather than the anatomical severity of the injuries. The RTS has been widely used in trauma centers, especially for triage purposes, as it can be quickly assessed in the pre-hospital setting. However, RTS does not account for the type, distribution, or severity of injuries, which can limit its ability to predict mortality in more complex trauma cases.

Trauma and Injury Severity Score (TRISS) The Trauma and Injury Severity Score (TRISS) combines the ISS (or NISS), the RTS, and the patient's age to estimate the probability of survival. TRISS has been widely validated and used in trauma registries as a comprehensive scoring system, considering both injury severity and physiological status. It has been shown to predict trauma-related mortality with good accuracy and is often used to assess trauma system performance and to guide clinical decision-making. However, TRISS may be less accurate in certain populations, such as older adults or those with significant comorbidities, as it primarily relies on injury-related factors and may not fully capture the complex interplay of clinical variables affecting outcomes.

Need for Comparative Studies While individual trauma scoring systems have demonstrated utility in predicting mortality, no single scoring system is universally superior. In clinical practice, there is a need to evaluate and compare these scoring systems across different populations and settings, particularly to determine which system is most reliable in predicting mortality for various trauma mechanisms.

injury patterns, and patient characteristics. Some studies have suggested that combining these systems may improve predictive accuracy, but evidence supporting the superiority of one over the others is inconclusive.

Additionally, while many studies have focused on the predictive validity of these scores in large datasets, fewer studies have compared them head-to-head within the same cohort of trauma patients. This gap in the literature necessitates a comprehensive, cohort-based study that directly compares the performance of the ISS, NISS, RTS, and TRISS for predicting mortality across a broad spectrum of trauma patients.

ELIGIBILITY:
Inclusion Criteria:

* Trauma patients admitted to the emergency room (ER).
* Documented injury data sufficient to calculate both the New Injury Severity Score (NISS) and the Injury Severity Score (ISS).
* Trauma scores (ISS, NISS, Revised Trauma Score [RTS], and Trauma and Injury Severity Score [TRISS]) calculated within 12 hour of arrival to ensure timely predictions.
* Informed consent provided by the patient or a legal guardian in cases of incapacity.

Exclusion Criteria:

* Under 18 years of age and pregnant women, due to differences in trauma management and scoring applicability.
* Non-trauma cases, including patients with terminal illnesses or severe cognitive impairments, to maintain focus on trauma outcomes.
* Incomplete trauma scoring, missing or incomplete medical records, and
* patients not treated in the trauma or emergency department.
* Patients who refuse participation or withdraw consent to ensure ethical participation.
* Transferred patients and those enrolled in other research studies that could interfere with trauma scoring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult trauma patients (≥18 years) presenting to the trauma and emergency department at Kadhimiya Educational Hospital in Baghdad. It includes individuals with acute injuries, such as blunt or penetrating trauma, who require trauma severity scoring. Data will be gathered through standardized clinical assessments and trauma scoring within the emergency department setting, ensuring a representative sample of the trauma population at the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
In hospital mortality | In-Hospital Phase (average of 7 days through discharge)
  Mortality (death) during hospitalization
Accuracy Assessment of Injury Severity Score (ISS) | the first 12 hours after ER admission
  Range: 0 to 75 Higher values indicate worse outcomes, reflecting greater injury severity.
Accuracy Assessment of New Injury Severity Score (NISS) | the first 12 hours after ER admission
  Range: 0 to 75. Higher values indicate worse outcomes, reflecting greater injury severity.
Accuracy Assessment of Trauma Injury Severity Score (TISS) | the first 12 hours after ER admission
  Range: 0 (represents a 0% probability of survival) to 1 (represents a 100% probability of survival), with higher scores indicating greater trauma severity.
Accuracy Assessment of the Revised Trauma Score (RTS) | the first 12 hours after ER admission
  The total RTS score ranges from 0 to approximately 12, with lower scores indicating more severe injuries and a higher risk of mortality.

SECONDARY OUTCOMES:
Length of Hospitalization | Up to discharge, an average of 7 days
  The total duration of a patient's stay in the hospital, measured from the date of admission to the date of discharge. This includes all days spent in general wards, intensive care units (ICU), and other hospital departments as part of their treatment course.
Number of Participants Requiring ICU Admission | Up to discharge, an average of 7 days
  The requirement for admission to the intensive care unit (ICU) is determined by the presence of severe clinical deterioration, significant complications, or the need for advanced monitoring and life-support measures.
Number of Participants Requiring Surgical Intervention | Up to discharge, an average of 7 days
  need for surgical intervention during a trauma patient's hospital stay.

CONTACTS AND LOCATIONS:
Locations (1):
- College of Medicine - Al-Nahrain University, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Senkowski CK, McKenney MG. Trauma scoring systems: a review. J Am Coll Surg. 1999 Nov;189(5):491-503. doi: 10.1016/s1072-7515(99)00190-8. No abstract available. PMID 10549738
- [Background] Champion HR, Sacco WJ, Copes WS, Gann DS, Gennarelli TA, Flanagan ME. A revision of the Trauma Score. J Trauma. 1989 May;29(5):623-9. doi: 10.1097/00005373-198905000-00017. PMID 2657085
- [Background] Baker SP, O'Neill B, Haddon W Jr, Long WB. The injury severity score: a method for describing patients with multiple injuries and evaluating emergency care. J Trauma. 1974 Mar;14(3):187-96. No abstract available. PMID 4814394
- [Result] Hoke MH, Usul E, Ozkan S. Comparison of Trauma Severity Scores (ISS, NISS, RTS, BIG Score, and TRISS) in Multiple Trauma Patients. J Trauma Nurs. 2021 Apr-Jun 01;28(2):100-106. doi: 10.1097/JTN.0000000000000567. PMID 33667204
- [Result] Boyd CR, Tolson MA, Copes WS. Evaluating trauma care: the TRISS method. Trauma Score and the Injury Severity Score. J Trauma. 1987 Apr;27(4):370-8. PMID 3106646
- [Result] Osler T, Baker SP, Long W. A modification of the injury severity score that both improves accuracy and simplifies scoring. J Trauma. 1997 Dec;43(6):922-5; discussion 925-6. doi: 10.1097/00005373-199712000-00009. PMID 9420106